CLINICAL TRIAL: NCT06222476
Title: A Multicentric, Prospective, Randomized Study Evaluating the Improvement of Renal Function Outcomes With Dorzagliatin in Patients With Type 2 Diabetes Mellitus With Early Kidney Injury.
Brief Title: Effect of Dorzagliatin on Renal Function Outcomes in People With Type 2 Diabetes: a Multicentric, Prospective, Randomized Study.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yan Bi (Other)
Responsible Party: Sponsor-Investigator, Yan Bi, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Organization: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BY2023
Record Dates: First submitted 2024-01-16; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Diabetic Nephropathy Type 2
MeSH Terms: interventions — Dorzagliatin; Gliclazide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients treat with Dorzagliatin (Experimental): Dorzagliatin will be initiated and maintained at 75mg twice a day until the completion of the study. Meanwhile, all patients will also continue on regimen of metformin 500mg three times a day throughout the study. Visits at 4-week intervals will be performed to evaluate the safety of drugs.
  Interventions: Drug: Dorzagliatin
- Patients treat with Gliclazide (Active Comparator): Gliclazide will be initiated and maintained at 30mg once a day until the completion of the study. Meanwhile, all patients will also continue on regimen of metformin 500mg three times a day throughout the study. Visits at 4-week intervals will be performed to evaluate the safety of drugs.
  Interventions: Drug: Gliclazide

INTERVENTIONS:
Drug: Dorzagliatin — Dorzagliatin will be initiated and maintained at 75mg twice a day
  Arms: Patients treat with Dorzagliatin
Drug: Gliclazide — Gliclazide will be initiated and maintained at 30mg once a day
  Arms: Patients treat with Gliclazide

SUMMARY:
The main purpose of this study is to explore the improvement of renal function before and after the intervention of dorzagliatin in patients with type 2 diabetes.

DETAILED DESCRIPTION:
As soon，metformin、SGLT-2i、GLP-1RA have been confirmed to have protective effect on the kidneys in the statement of consensus at home and abroad. Dorzagliatin exerts a potent hypoglycemic effect by activating glucokinase and is not affected by the patient's renal function. However, previous studies of this drug have rarely involved studies that improve markers related to renal function. On the one hand, in this study, changes of renal function (eGFR, creatinine, cystatin C, TNF-1) are collected to investigate whether dorzagliatin is benefit to kidney. On the other hand, renal magnetic resonance imaging(MRI) results are analysed to explore the differences among control subjects and patients treated with dorzagliatin.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-75 years old, male and female.
2. Patients with type 2 diabetes mellitus, type 2 diabetes mellitus diagnosis criteria: according to the "Chinese Type 2 Diabetes Mellitus Prevention and Treatment Guide (2020 Edition).
3. UACR 30-299mg/g.
4. eGFR ≥60mL/min/1.73m².
5. HbA1c 7.0-10.5%.

Exclusion Criteria:

1. Pregnant and lactating women and women of childbearing age who do not want to take reliable contraceptive measures.
2. Known allergic history to dorzagliatin/gliclazide/metformin.
3. Diabetic acute and chronic complications, including diabetic ketoacidosis, a hyperglycemic hyperosmolar state or hypoglycemic coma, etc.
4. Serious impairment of heart, liver, kidney and other organs.
5. With hypertension(≥140/90mmHg).
6. Fasting C-peptide <300pmol/L.
7. Contraindications of MRI examination, such as implantation of metal prosthesis in vivo, claustrophobia, wearing insulin pumps, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-02-20 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Participants' personal information | 1 day
  Self-reported information (age in years, gender，course of disease )
Physical assessments | 1 day
  BMI (body mass index) in kg/m^2
renal function | 1 day
  changes of renal function (eGFR, creatinine, cystatin C, TNF-1)
renal magnetic resonance imaging(MRI) | 1 day
  Changes of perirenal fat content, renal proton density fat fraction and degree of renal fibrosis

SECONDARY OUTCOMES:
blood sugar | 1 day
  fasting blood sugar、2-hour postprandial blood sugar
insulin | 1 day
  fasting insulin、2-hour insulin
HOMA2-β | 1 day
  20*fasting insulin（mIU/L）/（fasting blood sugar（mmol/L）-3.5）
HOMA2-IR | 1 day
  fasting blood sugar（mmol/L）*fasting insulin（mIU/L）/22.5
HOMA2-IS | 1 day
  22.5/fasting blood sugar（mmol/L）*fasting insulin（mIU/L）

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yang W, Zhu D, Gan S, Dong X, Su J, Li W, Jiang H, Zhao W, Yao M, Song W, Lu Y, Zhang X, Li H, Wang G, Qiu W, Yuan G, Ma J, Li W, Li Z, Wang X, Zeng J, Yang Z, Liu J, Liang Y, Lu S, Zhang H, Liu H, Liu P, Fan K, Jiang X, Li Y, Su Q, Ning T, Tan H, An Z, Jiang Z, Liu L, Zhou Z, Zhang Q, Li X, Shan Z, Xue Y, Mao H, Shi L, Ye S, Zhang X, Sun J, Li P, Yang T, Li F, Lin J, Zhang Z, Zhao Y, Li R, Guo X, Yao Q, Lu W, Qu S, Li H, Tan L, Wang W, Yao Y, Chen D, Li Y, Gao J, Hu W, Fei X, Wu T, Dong S, Jin W, Li C, Zhao D, Feng B, Zhao Y, Zhang Y, Li X, Chen L. Dorzagliatin add-on therapy to metformin in patients with type 2 diabetes: a randomized, double-blind, placebo-controlled phase 3 trial. Nat Med. 2022 May;28(5):974-981. doi: 10.1038/s41591-022-01803-5. Epub 2022 May 12. PMID 35551292
- [Background] Simons PIHG, Simons N, Stehouwer CDA, Schalkwijk CG, Schaper NC, Brouwers MCGJ. Association of common gene variants in glucokinase regulatory protein with cardiorenal disease: A systematic review and meta-analysis. PLoS One. 2018 Oct 23;13(10):e0206174. doi: 10.1371/journal.pone.0206174. eCollection 2018. PMID 30352097
- [Background] Hishida A, Takashima N, Turin TC, Kawai S, Wakai K, Hamajima N, Hosono S, Nishida Y, Suzuki S, Nakahata N, Mikami H, Ohnaka K, Matsui D, Katsuura-Kamano S, Kubo M, Tanaka H, Kita Y. GCK, GCKR polymorphisms and risk of chronic kidney disease in Japanese individuals: data from the J-MICC Study. J Nephrol. 2014 Apr;27(2):143-9. doi: 10.1007/s40620-013-0025-0. Epub 2013 Dec 17. PMID 24535998
- [Background] Wang K, Shi M, Yang A, Fan B, Tam CHT, Lau E, Luk AOY, Kong APS, Ma RCW, Chan JCN, Chow E. GCKR and GCK polymorphisms are associated with increased risk of end-stage kidney disease in Chinese patients with type 2 diabetes: The Hong Kong Diabetes Register (1995-2019). Diabetes Res Clin Pract. 2022 Nov;193:110118. doi: 10.1016/j.diabres.2022.110118. Epub 2022 Oct 13. PMID 36243233
- [Background] Lin L, Dekkers IA, Huang L, Tao Q, Paiman EHM, Bizino MB, Jazet IM, Lamb HJ. Renal sinus fat volume in type 2 diabetes mellitus is associated with glycated hemoglobin and metabolic risk factors. J Diabetes Complications. 2021 Sep;35(9):107973. doi: 10.1016/j.jdiacomp.2021.107973. Epub 2021 Jun 15. PMID 34217586